CLINICAL TRIAL: NCT07353437
Title: Fluzoparib as Adjuvant Treatment in Patients With Germline Homologous Recombination Repair (HRR) Mutated Primary Breast Cancer (Flamenco)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Keda Yu, chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Flamenco
Record Dates: First submitted 2026-01-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluzoparib group (Experimental)
  Interventions: Drug: Fluzoparib
- Physician choice (Active Comparator)
  Interventions: Drug: Physician choice

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib 100 mg bid for 1 year
  Arms: Fluzoparib group
Drug: Physician choice — Standard treatment chosen by physician (in case of TNBC, combination therapy includes but is not limited to immunotherapy or capecitabine; in case of HR +, combination therapy includes but is not limited to endocrine therapy or CDK4/6 inhibitors)
  Arms: Physician choice

SUMMARY:
The study is a randomized, open-label, multicenter phase II clinical trial of the efficacy and safety of fluzopanib in the adjuvant treatment of early breast cancer using germline mutations in homologous recombination repair pathway genes. Study design Patients will be randomized into 2 groups in a 1:1 ratio after enrollment:

Experimental group: fluzoparib, specific: fluzoparib 100 mg bid for 1 year. As well as the standard of care selected by the physician (in case of TNBC, combination therapy includes but is not limited to immunotherapy or capecitabine; in case of HR +, combination therapy includes but is not limited to endocrine therapy or CDK4/6 inhibitors).

Control group: Doctors' choice of standard treatment (in case of TNBC, combination therapy includes but is not limited to immunotherapy or capecitabine; in case of HR +, combination therapy includes but is not limited to endocrine therapy or CDK4/6 inhibitors)

ELIGIBILITY:
Inclusion Criteria:

* Female 18-75 years
* ECOG 0-1
* Histologically confirmed invasive carcinoma (regardless of pathological type)
* No gross or microscopic residual tumor after surgical resection
* For triple-negative early breast cancer receiving neoadjuvant therapy (at least 6 cycles of chemotherapy), postoperative pathological assessment of non-pCR is required; for ER and/or PgR-positive and HER2-negative early breast cancer receiving neoadjuvant therapy (at least 6 cycles of chemotherapy or endocrine therapy), postoperative pathological assessment of non-pCR and ypLN + is required; for triple-negative early breast cancer not receiving neoadjuvant therapy, postoperative pathological assessment of ≥ pT2 or ≥ pN1 is required; for ER and/or PgR-positive and HER2-negative early breast cancer not receiving neoadjuvant therapy, postoperative pathological assessment of ≥ 4 positive lymph nodes or 1-3 positive lymph nodes with high-risk factors (tumor diameter ≥ 5 cm, or histological grade 3, or Ki-67 ≥ 30%) is required
* Carrying pathogenic or possibly pathogenic mutations in BARD1/BRIP1/EXO1/FANCM/NBN/PALB2/PARP1/PARP2/POLQ/RAD50/RAD51/RAD51B/RAD51C/RAD51D/RAD52/RAD54L/RE/QL5/RFC1/RPA1/TOP3A/TOP3B/BLM germline genes confirmed by second-generation sequencing or first-generation sanger sequencing

Exclusion Criteria:

* Bilateral breast cancer or carcinoma in situ DCIS/LCIS;
* Metastases at any site;
* contralateral breast clinical or imaging suspected malignant but not confirmed, need biopsy;
* Treated for advanced disease;
* Patients who have received tamoxifen, raloxifene, or aromatase inhibitors (AIs) to reduce the risk of breast cancer ("chemoprevention") and/or who have previously undergone prophylactic ovariectomy within 2 years;
* Malignant tumor (except skin basal cell carcinoma and cervical carcinoma in situ) within 5 years, including contralateral breast cancer;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
iDFS | 3-year iDFS
  DFS, Invasive Disease-Free Survival, refers to the time from randomization to the first occurrence of locoregional invasive recurrence, distant metastasis, contralateral invasive tumor, or death from any cause. The primary endpoint of this study is 3-year iDFS.

IPD SHARING:
Plan to Share IPD: No